CLINICAL TRIAL: NCT05676008
Title: A Study of Positive Emotions With Long COVID (Post-Acute Sequelae of SARS CoV-2 Infection)
Brief Title: A Study of Positive Emotions With Long COVID-19
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1840049
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: Mindfulness
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control (No Intervention)
- Treatment (Experimental)
  Interventions: Behavioral: Microdosing of mindfulness

INTERVENTIONS:
Behavioral: Microdosing of mindfulness — The intervention consists of two parts: 1) four structured training sessions offered as online synchronous classes, and 2) self-microdosing of mindfulness activities in everyday life.
  Arms: Treatment

SUMMARY:
This study is testing a new brief mindfulness practice for people suffering from long COVID-19 symptoms. People suffering from long COVID are particularly vulnerable to negative emotions, as they must also cope with the long-term uncertainty of physical and psychological stress beyond the acute infection. The goal of the study is to measure the ability of a brief mindfulness practice to promote a sense of well-being in people suffering from long COVID.

DETAILED DESCRIPTION:
This is a pilot randomized waitlist-controlled clinical trial (RCT) testing a new brief self-care intervention for people suffering from post-acute sequelae SARS-CoV-2 infection (PASC). The overarching goal of this study is to establish the feasibility and early efficacy of microdosing mindfulness as a self-care intervention. The purpose of the intervention is to promote a sense of well-being among PASC patients who currently have limited access to other proven self-care modalities.

Our research question is whether our newly developed training can assist PASC patients to self-microdose mindfulness (5-15 seconds activities in everyday life) and improve on perceived metrics of well-being (primary outcome). Our hypothesis is that self-microdosing mindfulness will evoke positive emotions that can improve well-being on patients suffering of PASC-related symptoms beyond 3 months post COVID-19 infection. If effective, an increased frequency of the mindfulness activity will then help buffer negative emotions (e.g., anger, loneliness, etc.) experienced during the pandemic and associated with ongoing stress and/or somatic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Able to participate in online zoom sessions and complete online surveys for 3 months
* English speakers
* Had a mild to moderate in severity COVID-19 infection > 3 months ago, feeling unwell, and are still experiencing in the present at least one PASC-related symptoms:
* Coughing or feeling short of breath
* Loss of smell or change in taste
* Recurrent Fever
* Body aches, headaches, chest pain, or stomach pain
* Brain fog (feeling like you can't think clearly)
* Having trouble sleeping
* Feeling very tired
* Mood changes

Exclusion Criteria:

* Adults that were admitted to an intensive care unit or placed on a respirator, had invasive heart (heart catheterization) or lung tests (bronchoscopy) performed.
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Well-being | 1 month
  14 items from the Mental Health Continuum Short Form

SECONDARY OUTCOMES:
Perceived Stress | 1, 3 and 12 months
  Perceived Stress Scale
Anxiety symptoms | 1, 3 and 12 months
  Generalized Anxiety Disorder scale
Depressive symptoms | 1, 3 and 12 months
  Beck Depression Inventory Short Form
Physical health | 1, 3 and 12 months
  Physical health symptoms - 11 items + 3 items of COVID symptoms
Cardiac symptoms | 1, 3 and 12 months
  Cardiac symptoms by the Kansas City Cardiomyopathy Questionnaire-12 items (KCCQ-12)
Well-being | 3 and 12 months
  14 items from the Mental Health Continuum Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Javier E Lopez, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monroy M, Amster M, Eagle J, Zerwas FK, Keltner D, Lopez JE. Awe reduces depressive symptoms and improves well-being in a randomized-controlled clinical trial. Sci Rep. 2025 May 12;15(1):16453. doi: 10.1038/s41598-025-96555-w. PMID 40355653